CLINICAL TRIAL: NCT03351868
Title: Gene Transfer for Fanconi Anemia Using a Self-inactivating Lentiviral Vector
Brief Title: FANCA Gene Transfer for Fanconi Anemia Using a High-safety, High-efficiency, Self-inactivating Lentiviral Vector
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17021
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Fanconi Anemia
Keywords: Fanconi anemia; Lentiviral vector; FANCA; Gene
MeSH Terms: conditions — Fanconi Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gene-modified autologous stem cells (Experimental): Autologous hematopoeitic stem cells and mesenchymal stem cells transduced with lentiviral vector carrying the FANCA gene ex vivo
  Interventions: Genetic: Gene-modified autologous stem cells

INTERVENTIONS:
Genetic: Gene-modified autologous stem cells — Infusion for 5x10^6~1x10^7 per kilogram of body weight of gene-modified cells; or more infusions depending on the circumstances

SUMMARY:
This is a Phase I/II clinical trial of gene therapy for treating Fanconi anemia using a self-inactivating lentiviral vector to functionally correct the defective gene. The objectives are to evaluate the safety and efficacy of the gene transfer clinical protocol.

DETAILED DESCRIPTION:
Fanconi anemia is a rare, inherited disease that is caused by a gene defect and that primarily affects an individual's bone marrow, resulting in decreased production of blood cells. The major problem for most patients is aplastic anemia, the blood counts for red blood cells, white blood cells, and platelets are low. In addition, some patients have physical defects usually involving the skeleton and kidneys. Fanconi anemia is typically diagnosed in childhood, and there is a high fatality rate. Hematopoietic stem cell transplantation (HSCT) is a common treatment for Fanconi anemia. However, there are many risks associated with HSCT including rejection of the transplanted cells and graft-versus-host disease.

The primary objectives are to evaluate the safety of the self-inactivating lentiviral vector, the ex vivo gene transfer clinical protocol and the efficacy of immune reconstitution in patients overcoming immune abnormalities present at the time of treatment, assessment of gene correction efficiency, and finally the long-term correction of Fanconi anemia associated disease symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Fanconi anemia FANCA type based on DNA sequencing and sensitivity test for chromosomal cleavage by mitomycin C or butylene oxide.
2. No cytogenetic abnormalities and the proportion of myelodysplastic abnormalities does not exceed 5% within 3 months prior to stem cell collection.
3. Age: ≥ 4 years.
4. Karnofsky: ≥ 70%.
5. ANC ≥ 5×10^8/L; PLT ≥ 2×10^10/L.
6. Hemoglobin ≥ 8g/dL.
7. Proper renal and hepatic functions (ULN denotes "upper limit of normal range") with

   * serum creatinine ≤ 1.5×ULN;
   * serum bilirubin ≤ 3×ULN;
   * AST/ALT ≤ 5×ULN.
8. Pulmonary function is normal; DLCO > 50%.
9. Written, informed consent obtained prior to any study-specific procedures.

Exclusion Criteria:

1. Diagnosis of active malignant disease or myelodysplastic syndrome.
2. Diagnosis of myeloid leukemia.
3. Pregnant or lactating females.
4. Existence of an available HLA-identical related donor.
5. Subject infected with HBV (HBsAg positive), HIV (HIV antibody positive), HTLV (HTLV antibody positive), Treponema pallidum antibody positive or TB culture positive.
6. Patients, in the opinion of investigators, may not be eligible or not able to comply with the study.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety in patients using CTCAE version 4.0 standard to evaluate the level of adverse events | 6 months
  Physiological parameter (measuring cytokine response, fever, symptoms)

SECONDARY OUTCOMES:
Treatment responses | 1 year
  Blood routine indexes will be obtained before and after treatment. Objective response, such as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria
Quality of life | 1 year
  Quality of life will be measured using the Functional Assessment of Cancer Therapy-General (FACT-G) before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, Ph.D, Principal Investigator — Shenzhen Geno-Immune Medical Institute; Xiao-Dong Shi, M.D./Ph. D, Study Director — Capital Institute of Pediatrics affiliated Children's hospital; Jie Zheng, M.D./Ph. D, Study Director — Beijing Children's Hospital
Locations (3):
- China (3):
  - Capital Institute of Pediatrics affiliated Children's hospital, Beijing, Beijing Municipality
  - Beijing Children's Hospital, Beijing, Beijing Municipality
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No